CLINICAL TRIAL: NCT02475629
Title: A Phase 3, Single Arm, 24-Week, Multicenter Study of Ibalizumab Plus an Optimized Background Regimen (OBR) in Treatment-Experienced Patients Infected With Multi-Drug Resistant HIV-1
Brief Title: Ibalizumab Plus Optimized Background Regimen in Patient With Multi-Drug Resistant HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMB-301
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-02

CONDITIONS: HIV
MeSH Terms: interventions — ibalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Ibalizumab plus OBR (Experimental): 2000 mg intravenous ibalizumab (loading dose) on Day 7 followed in 14 days (on Day 21) by 800 mg intravenous ibalizumab administered once every two weeks, plus an Optimized Background Regimen (OBR) beginning on Day 14.
  Interventions: Biological: ibalizumab; Drug: Optimized Background Regimen (OBR)

INTERVENTIONS:
Biological: ibalizumab — 2000mg intravenous ibalizumab (loading dose), followed 14 days later by 800mg intravenous ibalizumab every 2 weeks
  Other Names: TNX-355; Hu1A8
Drug: Optimized Background Regimen (OBR) — All participants will be prescribed an Optimized Background Regimen of antiretroviral medications selected on the basis of treatment history and the results of Screening viral resistance and tropism testing. The prescribed regimen must contain at least one agent to which the participant's virus is known to be sensitive.

SUMMARY:
This Phase 3, single arm, multicenter study will evaluate the safety and effectiveness of ibalizumab in treatment-experienced patients infected with multi-drug resistant HIV-1.

DETAILED DESCRIPTION:
This Phase 3, single arm, multicenter study will evaluate the safety and effectiveness of ibalizumab in treatment-experienced patients infected with multi-drug resistant HIV-1. Patients must have been treated with HAART for at least 6 months and be failing or have recently failed (i.e., in the last 8 weeks) therapy to determine baseline viral load.

Days 0-6 of the study will be a "control period." During Days 0 through 6 patients will be monitored on current failing therapy (or no therapy, if the patient has failed and discontinued treatment within the 8 weeks preceding Screening).

Days 7-13 of the study will be an "essential monotherapy period." During Days 7 through 13 patients will continue on current failing therapy and receive one 2000 mg dose (loading dose) of ibalizumab on Day 7. Day 7 is Baseline for the treatment period (Day 7-Week 25).

Day 14-Week 25 of the study will be the "maintenance period." On Day 14 (primary endpoint), the OBR will be initiated and must include at least one agent to which the patient's virus is susceptible. Beginning at Day 21, 800 mg of ibalizumab will be administered every 2 weeks through Week 23.

End of Study evaluations will be performed at Week 25, and a follow-up visit will be conducted at Week 29.

ELIGIBILITY:
Inclusion Criteria:

* Are capable of understanding and have voluntarily signed the informed consent document
* Have documented HIV-1 infection by official, signed, written history (e.g., laboratory report), otherwise an HIV-antibody test will be performed
* Have no acquired immunodeficiency syndrome (AIDS)-defining events in the 3 months before Screening, other than cutaneous Kaposi's sarcoma or wasting syndrome due to HIV
* Are able and willing to comply with all protocol requirements and procedures
* Have a life expectancy that is >6 months.
* Have a viral load >1,000 copies/mL and documented resistance to at least one antiretroviral medication from each of three classes of antiretroviral medications as measured by resistance testing
* Have a history of at least 6 months on antiretroviral treatment
* Are receiving a stable highly active antiretroviral regimen for at least 8 weeks before Screening and are willing to continue that regimen until Day 14, OR (in the past 8 weeks) have failed and are off therapy and are willing to stay off therapy until Day 14
* Have full viral sensitivity/susceptibility to at least one antiretroviral agent, other than ibalizumab, as determined by the screening resistance tests and be willing and able to be treated with at least one agent to which the patient's viral isolate is fully sensitive/susceptible according to the screening resistance tests as a component of OBR
* If sexually active, are willing to use an effective method of contraception during the study and for 30 days after the last administration of the study drug

Exclusion Criteria:

* Any active AIDS-defining illness per Category C conditions according to the Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection, with the following exceptions: cutaneous Kaposi's sarcoma and wasting syndrome due to HIV
* Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined from screening, medical history and/or physical examination that, in the investigator's opinion, would preclude the patient from participating in this study
* Any significant acute illness within 1 week before the initial administration of study drug
* Any active infection secondary to HIV requiring acute therapy; however, patients that require maintenance therapy (i.e., secondary prophylaxis for opportunistic infections) will be eligible for the study.
* Any immunomodulating therapy (including interferon), systemic steroids, or systemic chemotherapy within 12 weeks before Enrollment
* Any prior exposure to ibalizumab (formerly TNX-355 and Hu5A8)
* Any vaccination within 7 days before Enrollment
* Any female patient who either is pregnant, intends to become pregnant, or is currently breastfeeding
* Any current alcohol or illicit drug use that, in the investigator's opinion, will interfere with the patient's ability to comply with the study schedule and protocol evaluations
* Any previous clinically significant allergy or hypersensitivity to any excipient in the ibalizumab formulation
* Any radiation therapy during the 28 days before first administration of investigational medication
* Any Grade 3 or 4 laboratory abnormality according to the Division of AIDS grading scale, except for the following asymptomatic Grade 3 events triglyceride elevation total cholesterol elevation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (27):
  - Long Beach Education and Research Consultants, Long Beach, California
  - W King Health Care Group, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Ruane Medical and Clinical Research Institute, Los Angeles, California
  - Charles R. Drew Univ. of Med. & Science Clinical and Translational Research Center, Los Angeles, California
  - Anthony Mills, MD, Inc., Los Angeles, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Palmtree Clinical Research Inc., Palm Springs, California
  - Quest Clinical Research, San Francisco, California
  - Kaiser Foundation Research Institute, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Circle Care Center, LLC, Norwalk, Connecticut
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute, West Palm Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Henry Ford Health Systems, Detroit, Michigan
  - St. John Hospital and Medical Center, Southfield, Michigan
  - ACRIA, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - Research Access Network, Houston, Texas
- Clinical Research PR, Inc, San Juan, Puerto Rico
- Taiwan (2):
  - E-Da Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Emu B, Fessel J, Schrader S, Kumar P, Richmond G, Win S, Weinheimer S, Marsolais C, Lewis S. Phase 3 Study of Ibalizumab for Multidrug-Resistant HIV-1. N Engl J Med. 2018 Aug 16;379(7):645-654. doi: 10.1056/NEJMoa1711460. PMID 30110589

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-Label Ibalizumab Plus OBR
Started | 40
Completed | 31
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Death | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Subject non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2
  United States | 34
  Taiwan | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Proportion of Participants Achieving a Viral Load Reduction of at Least 0.5 Log 10: ITT-MEF
Description: Proportion of participants (%) achieving a viral load reduction of at least 0.5 log from baseline (Day 7)
Time Frame: Day 14
Population: Intent to Treat (ITT) Population (all participants enrolled) with missing values set to zero change
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
proportion of participants | 0.825 [0.6772 to 0.9266]

2. Primary Outcome: Efficacy: Proportion of Subjects With a Viral Load Decrease of at Least 0.5 Log 10 - Protocol Correct
Description: Proportion of patients (%) with a viral load decrease of at least 0.5 log 10 from baseline (day 7)
Time Frame: Day 14
Population: Protocol Correct (PC) Population (all participants with non-missing viral load assessments at Day 7, Day 14 and Week 25/End of Study)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 26
proportion of participants | 0.846 [0.6513 to 0.9564]

3. Secondary Outcome: Efficacy: Proportion of Patients With Undetectable Viral Load: ITT-MEF
Description: Proportion of patients with undetectable Viral Load (<50 copies/mL, and <400 copies/mL)
Time Frame: Week 25 /end of study
Population: Intent to Treat (ITT) Population (all participants enrolled) with missing values set to failure
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
proportion of participants
  <50 copies/mL | .425 [0.2704 to 0.5911]
  <400 copies/mL | .525 [0.3613 to 0.6849]

4. Secondary Outcome: Efficacy: Proportion of Patients With Undetectable HIV-RNA Levels: Protocol Correct
Description: Proportion of patients (%) with HIV-RNA levels < 50 copies/mL and < 400 copies/mL at Week 25/End of Study
Time Frame: Week 25/End of Study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 26
proportion of participants
  <50 copies/mL | .654 [0.4433 to 0.8279]
  <400 copies/mL | .808 [0.6065 to 0.9345]

5. Secondary Outcome: Mean Change in Viral Load as a Measure of Efficacy - ITT-MEF
Description: Mean change from Day 7/Baseline in log 10 vial load measured at Day 14
Time Frame: Day 7 and Day 14
Population: Intent to Treat (ITT) Population (all participants enrolled) with missing values set to zero change
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Log10 copies/mL | -1.07 (0.618)

6. Secondary Outcome: Mean Change in Viral Load as a Measure of Efficacy - Protocol Correct
Description: Mean change from Day 7/Baseline in Log 10 viral load measured at Day 14
Time Frame: Day 7 and Day 14
Population: Protocol Correct (PC) Population (all participants with non-missing viral load assessments at Day 14
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 26
Log10 copies/mL | -1.11 (0.641)

7. Secondary Outcome: End of Study Viral Load Reductions as a Measure of Efficacy - Intent to Treat Analysis
Description: Proportion of patients achieving a >/= 0.5 log10 and >/= 1.0 log10 decrease from Day 7/Baseline in viral load at Week 25/End of Study
Time Frame: at Week 25/End of Study
Population: Intent to Treat (ITT) Population (all participants enrolled) with missing values set to zero change
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
proportion of participants
  >/= 0.5 log10 reduction | .625 [0.4580 to 0.7727]
  >/= 1.0 log10 reduction | .550 [0.3849 to 0.7074]

8. Secondary Outcome: End of Study Viral Load Reductions as a Measure of Efficacy - Protocol Correct Analysis
Description: as for outcome 7
Time Frame: at Week 25/End of Study
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 26
proportion of participants
  >/= 0.5 log10 reduction | .962 [0.8036 to 0.9990]
  >/= 1.0 log10 reduction | .846 [0.6513 to 0.9564]

9. Secondary Outcome: Mean Change in CD4+ Cell Count as a Measure of Efficacy and Safety - ITT
Description: Mean change from Day 7/Baseline in CD4+ cell count at Week 25/End of Study
Time Frame: Day 7 and Week 25/End of Study
Population: Intent to Treat (ITT) Population (all participants enrolled). Only obtained values were included in analysis - missing values were not imputed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 27
cells/mm^3 | 62.4 (105.75)

10. Secondary Outcome: Mean Change in CD4+ Cell Count as a Measure of Efficacy and Safety - Protocol Correct
Description: Mean change from Day 7/Baseline in CD4+ cell count at Week 25/End of Study
Time Frame: Day 7 and Week 25/End of Study
Population: Protocol Correct (PC) Population (all participants with non-missing viral load assessments at Day 7, Day 14 and Week 25/End of Study) with non-missing CD4+ cell count measurements
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 22
cells/mm^3 | 67.0 (114.35)

11. Secondary Outcome: Safety: Proportion of Participants Experiencing Adverse Events
Description: Proportion of participants experiencing at least one treatment emergent adverse event to week 25/End of Study
Time Frame: Through Week 25/End of Study
Population: All participants receiving at least one partial dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Participants | 32

12. Secondary Outcome: Proportion of Participants Experiencing Adverse Event Related to Study Drug as a Measure of Safety and Tolerability
Description: Proportion of participants experiencing a treatment emergent adverse event determined by the investigator to be related to study drug
Time Frame: Through Week 25/End of Study
Population: All participants receiving at least one partial dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Participants | 7

13. Secondary Outcome: Proportion of Participants Experiencing Serious Adverse Event as a Measure of Safety and Tolerability
Description: Proportion of participants experiencing at least one serious treatment emergent adverse event, excluding death
Time Frame: Through Week 25/End of Study
Population: All participants receiving at least one partial dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Participants | 9

14. Secondary Outcome: Proportion of Participants Discontinuing Study Drug Due to Adverse Event
Description: Proportion of participants discontinuing study drug due to occurrence of treatment emergent adverse event
Time Frame: Through Week 25/End of Study
Population: All participants receiving at least one partial dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Participants | 5

15. Secondary Outcome: Proportion of Participants Experiencing Adverse Event Grade 3 and Higher as a Measure of Safety and Tolerability
Description: Proportion of participants experiencing treatment emergent adverse event Grade 3 and higher
Time Frame: Through Week 25/End of Study
Population: All participants receiving at least one partial dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Participants | 11

16. Secondary Outcome: Proportion of Participants Experiencing Adverse Event With Death as Outcome as a Measure of Safety and Tolerability
Description: Proportion of participants experiencing treatment emergent adverse event with death as the outcome, regardless of relationship to study drug
Time Frame: Through Week 25/End of Study
Population: All participants receiving at least one partial dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Participants | 4

17. Secondary Outcome: Proportion of Participants Experiencing New AIDS-defining Adverse Event According to CDC Criteria as a Measure of Safety and Tolerability
Description: Proportion of participants experiencing treatment emergent adverse event that is AIDS-defining by the CDC adverse event classification criteria for HIV infection
Time Frame: Through Week 25/End of Study
Population: All participants receiving at least one partial dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 40
Participants | 4

18. Other Pre Specified Outcome: Pharmacodynamics: CD4 Receptor Occupancy
Description: % of CD receptors occupied by ibalizumab on CD4+ T-cells
Time Frame: At Week 25/End of Study
Population: Intent to Treat (ITT) Population (all participants enrolled) with non-missing receptor occupancy assessments
Measure: Mean (Standard Deviation); unit: percentage of receptors
Arm/Group | Open-Label Ibalizumab Plus OBR
Number analyzed (Participants) | 27
percentage of receptors | 90.40 (32.909)

ADVERSE EVENTS:
Time Frame: Through Week 29
Description: At every participants were asked a nondirective question to elicit any medically related changes, including whether they had been hospitalized, had any accidents, used any new medications, or changed concomitant medication. AEs also were documented from clinically significant findings resulting from abnormal laboratory test values, physical examination findings, ECG abnormalities, or from other documents relevant to safety.
Arm/Group | Open-Label Ibalizumab Plus OBR
All-Cause Mortality (participants affected / at risk) | 4/40
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 32/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Ibalizumab Plus OBR (N=40)
Pyrexia (General disorders) | 2 (3)
Asthenia (General disorders) | 1 (2)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1)
Immune reconstitution inflammatory disorder (Immune system disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Ibalizumab Plus OBR (N=40)
Nasopharyngitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (15)
Nausea (Gastrointestinal disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 5 (6)
Pyrexia (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (12) — Rash is a combined count of all types of rashes reported, including rash, rash erythematous, rash generalised,rash macular, rash maculo-papular, rash papular, rash pruritic. No rash type occurred at a rate >/= 5%.
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No